CLINICAL TRIAL: NCT01476930
Title: Cupping Therapy and SERKANGABIN Versus Conventional Treatment of Migraine Headache: a Randomized Controlled Trial
Brief Title: Cupping and Serkangabin Versus Conventional Migraine Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Birjand University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: n231; n231hej (Other Grant/Funding Number: birjand university of medical sciences)
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Migraine Headache
Keywords: migraine; prophylactic treatment; cupping; serkangabin
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cupping serkangabin (Experimental): migraine cases treated by cupping and serkangabin syrup
  Interventions: Procedure: cupping and serkangabin syrup
- conventional (Active Comparator): migraine cases treated by conventional drug treatment protocols
  Interventions: Drug: conventional migraine drug treatment

INTERVENTIONS:
Procedure: cupping and serkangabin syrup — wet cupping serkangabin syrup
  Arms: cupping serkangabin
Drug: conventional migraine drug treatment — nortriptyline ,propranolol ,ergotamine , sumatriptan tablets
  Arms: conventional

SUMMARY:
Migraine is the most common recurrent headache. Current therapy of migraine headache consists of multiple drug groups for control of attack and prophylaxis against recurrent attacks. Emerging alternative medicine worldwide led investigators to evaluate the efficacy of cupping therapy plus SERKANGABIN syrup in treatment of migraine headache. Severity, duration and frequency of attacks of migraine headache evaluated in two groups during six months from presentation.

DETAILED DESCRIPTION:
In a randomized controlled trial investigators randomly assigned 76 patients with migraine to cupping therapy plus SERKANGABIN or to receive conventional medical treatment. The use of CAM in migraine is a growing phenomenon. Migraine patients seek and explore both conventional and CAM approaches. Wet cupping is an ancient medical technique still used in several contemporary societies. It is being used in management of hypertension, diabetes mellitus, and headaches, renal and biliary stones and for maintaining health. Little experimental study has been devoted to test its efficacy to treat migraine headache. Investigators planned this study for evaluation of therapeutic efficacy of wet cupping and an Iranian traditional medicine preparation, SERKANGABIN in treatment of migraine headache compared with current medicine protocols. SERKANGABIN is a preparation of honey, vinegar and distilled mint water that in traditional Iranian medicine is believed to have therapeutic effects in many diseases (diabetes mellitus, hypertension, hyperlipidemia, osteoarthritis, chronic obstructive airway disease, interstitial lung disease, hepatitis, fatty liver, ischemic heart disease, migraine, cerebrovascular diseases)

ELIGIBILITY:
Inclusion Criteria:

* migraine headache with or without aura

Exclusion Criteria:

* uncontrolled hypertension
* ischemic heart disease
* cardiac arrhythmia or symptomatic Wolff-Parkinson-White syndrome
* previous stroke or transient ischemic attack
* severe liver or renal impairment
* any other severe or disabling medical condition
* history of alcohol or analgesic or psychotropic drug abuse
* contraindication to or known hypersensitivity to study drugs
* current use or use in the previous 2 weeks of MAO-inhibitors
* a pain disorder other than migraine as the primary presenting problem
* current psychological treatment, psychiatric disorder needing immediate or priority treatment
* current or planned breast feeding or pregnancy or unwillingness to use an established contraceptive method
* non compliance of patients
* not presenting at times determined for treatment and evaluation

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 391 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
frequency of migraine attacks per week | 2 weeks after first presentation
  endpoints evaluated in both study groups 2 weeks after first presentation and receiving treatment protocols

SECONDARY OUTCOMES:
severity of migraine attacks | 2 weeks after first presentation
  severity of migraine attacks evaluated 2 weeks after first presentation in two study groups
duration of migraine attacks | 2 weeks after first presentation
  duration of migraine attacks evaluated 2 weeks after first presentationin two study groups
severity of migraine attacks | 1 month after first presentation
  severity of migraine attacks evaluated 1 month after first presentation in two study groups
severity of migraine attacks | 3 months after first presentation
  severity of migraine attacks evaluated 3 months after first presentation in two study groups
severity of migraine attacks | 6 months after first presentation
  severity of migraine attacks evaluated 6 months after first presentation in two study groups
duration of migraine attacks | 1 month after first presentation
  duration of migraine attacks evaluated 1 month after first presentation in two study groups
duration of migraine attacks | 3 months after first presentation
  duration of migraine attacks evaluated 3 months after first presentation in two study groups
duration of migraine attacks | 6 months after first presentation
  duration of migraine attacks evaluated 6 months after first presentation in two study groups
frequency of migraine attacks | 1 month after first presentation
  frequency of migraine attacks evaluated 1 month after first presentation in two study groups
frequency of migraine attacks | 3 months after first presentation
  frequency of migraine attacks evaluated 3 months after first presentation in two study groups
frequency of migraine attacks | 6 months after first presentation
  frequency of migraine attacks evaluated 6 months after first presentation in two study groups

CONTACTS AND LOCATIONS:
Overall Officials: mohammad khodashenas roudsari, M.D., Study Chair — assistant proffessor of internal medicine
Locations (1):
- Birjand University of Medical Sciences,Valiasr Hospital, Birjand, South Khorasan Province, Iran